CLINICAL TRIAL: NCT05573776
Title: A Pilot Study of the Effect of High Protein Supplement and Exercise Therapy on Preservation of Skeletal Muscle Mass and Quality of Life in Patients With Gastric Cancer and Pancreatic Cancer Treated With Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 4-2020-0455
Record Dates: First submitted 2022-09-26; First posted 2022-10-10 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Gastric Cancer; Pancreatic Cancer
MeSH Terms: conditions — Stomach Neoplasms; Pancreatic Neoplasms | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Therapy, High Protein supplement (Experimental)
  Interventions: Other: Exercise Therapy, High Protein supplement

INTERVENTIONS:
Other: Exercise Therapy, High Protein supplement — patients with gastric and pancreatic cancer will be eligible, and 30 patients will be randomly assigned to the exercise therapy + high protein supplement group and 30 patients to the exercise therapy + placebo supplement group.

SUMMARY:
For gastric and pancreatic cancer patients scheduled for primary chemotherapy, we would like to report muscle mass preservation and improvement in quality of life in Chinese characters that received only exercise therapy and high protein supplements at the same time

DETAILED DESCRIPTION:
Sixty patients with gastric and pancreatic cancer will be eligible, and 30 patients will be randomly assigned to the exercise therapy + high protein supplement group and 30 patients to the exercise therapy + placebo supplement group.

ELIGIBILITY:
Inclusion Criteria:

1. Has provided signed written informed Consent
2. Has a histologically confirmed gastric or pancreatic cancer
3. Has a patient scheduled for chemotherapy - Patients who are scheduled to be treated with TS-1 or Xelox for gastric cancer-adjuvant chemotherapy - Patients scheduled for primary chemotherapy for pancreatic cancer-progressive/transitional diseases

Exclusion Criteria:

1. Age under 19 or over 90 year of age
2. Eastern Cooperative Oncology Group (ECOG) ≥ 2
3. Patients with severe malnutritional evaluation (PG-SGAC)
4. Any of the following within 3 months prior to study recruitment: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, NYHA class III or IV congestive heart failure, stroke or transient ischemic attack.
5. A person with previous uncontrolled seizures, central nervous system or psychological disorders
6. Have uncontrolled active infection or sepsis
7. Have deep vein thrombosis occurs within 4 weeks prior to the start of test recruitment
8. Severe acute or chronic conditions that may reduce the patient's ability to participate in clinical trials or make it difficult to interpret clinical trial results
9. Pregnant or lactating women. Pregnancy test results are positive in childbearing women
10. Gastrointestinal obstruction, malabsorption syndrome, or diseases that significantly affect digestive functions

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Comparison of muscle mass between exercise therapy alone and high protein supplement combination groups | 6weeks
  Comparison of muscle mass between the exercise therapy single group and the high-protein supplement combination group as assessed by Bioelectrical impedance analsis (BIA) (performed in Week 6)
Comparison of muscle variation between exercise therapy alone and high protein supplement combination groups | 6weeks
  Comparison of muscle variation between the exercise therapy single group and the high-protein supplement combination group as assessed by Bioelectrical impedance analsis (BIA) (performed in Week 6)

SECONDARY OUTCOMES:
Exercise Compliance | 3years
  As assessed by compliance for planned exercise (aerobic/strength exercise) adherence rate (%)
High Protein/Placebo Supplement rate | 3years
  As assessed by compliance for planned high protein/placebo supplementation rate (%)
Quality of Life (QoL) Evaluation (Korean version EORTC QLQ-C30) | 3years
  European Organization for Research and Treatment Core Quality of Life Questionnaire (EORTC QLQ-C30) Korean version EORTC QLQ-C30 consists of 30 questions, and total score will be reported. Response options for each EPIC question form a Likert scale, and multi-item scale scores will be summed and transformed linearly to a 0-to-100 scale.
  The higher the score, the higher the quality of life. Using the QOL questionnaire (EOGRTC QLQ-C30), a total of 3 measurements were taken before chemotherapy and 1 week after chemotherapy.
Nutritional status assessment | 3years
  Nutritional status assessment for the exercise therapy single group versus the high-protein supplement combination group as assessed by PG-SGA(the Scored Patient-Generated Subjective Global Assessment)
Progression-free survival (PFS) | 3years
  Progression-free survival (PFS): To evaluate the treatment effect of High Protein/Placebo Supplement on progression-free survival (PFS) rate at 3years
Overall Survival (OS) | 3years
  Overall Survival (OS): The time from the date of first dose and the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Minkyu Jung, Principal Investigator — Yonsei Cancer Center, Yonsei University College of Medicine
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No